CLINICAL TRIAL: NCT06440200
Title: Applying Group Game-based Activities to Improve the Health of Patients With Chronic Mental Illness
Brief Title: Exploring the Health Effects of Group Game-based Activities on Individuals With Chronic Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202401209RINE
Record Dates: First submitted 2024-03-28; First posted 2024-06-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Chronic Mental Illness; Schizophrenia; Psychiatry
Keywords: group game-based activities; physiological values; depression rating scales; quality of life
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group gamed-based activites (Experimental): The group game-based activity will be twice a week lasting 12 weeks. There will be many motion sensing games in the group game-based activities. The games designed for activities can provide somatosensory control and visual and auditory feedback.
  Interventions: Behavioral: group gamed-based activity
- control group (No Intervention): The activities will be the psychiatric day wards and half-way house offered as usual.

INTERVENTIONS:
Behavioral: group gamed-based activity — Participants in interventional group will play the active-type software with Switch game console which develops by Nintendo company. Team building, cooperation, cohesion, sense of belonging and sense of achieving will be emphasized.
  Arms: group gamed-based activites

SUMMARY:
This study aims to explore the health effects of group games for patients with chronic mental illness. The goal of this clinical intervention study is to compare the efficacy of group games in two ways (experimental group/ group game-based or control group) to improve the health of patients with chronic mental illness. The main questions it aims to answer are:

The efficacy of applying group game-based activities to increase interest and improve the physical fitness of patients with chronic mental illness. Also, the goal of this clinical interventional study is to clarify the positive benefits of psychological and social aspects.

Subjects will be asked to complete the questionnaire and physical ability examination after filling out the consent of this study. Participants will be randomly divided into two groups. Participants in the experimental group will accept the group game-based activities for 12 weeks (twice per week, 22 times). In contrast, Participants in the control group will accept the activities the psychiatric day wards and halfway house offer as usual. After 12 weeks of intervention, The Participants in both groups will be asked to fill out the questionnaire and physical ability examination. One month later, Participants in both groups will be asked to fill out the questionnaire and physical ability examination again. The study will last for 4 months. The time points for completing the questionnaire are listed following:

Baseline/ pre-intervention test(T1), First post-intervention test (T2, 12 weeks later) and Second post-intervention test (T3, 4 weeks later). The researchers will compare the difference in effectiveness between the two groups.

DETAILED DESCRIPTION:
This study is a randomized controlled study. Researchers use a random assignment. One is an experimental group (group game-based), and the other is a control group(activities as usual). This Parallel two-group pre-test, first post-test and second post-test are designed to conduct a 12-week interventional study regarding group game-based activities for patients with chronic mental illness. A total of 3 questionnaires will be collected to compare the differences between the two groups to clarify the efficacy of group game-based activities. The investigators will discuss the outcome and the change in physiological values, physical ability, depression rating scale, quality of life and the motivation of group game-based activities.

Once the participants fill out the consent form, they will be asked to conduct the pre-test questionnaire including physiological values, physical ability, depression rating scale and quality of life. Then, the random numbers table will be used to divide subjects into the experimental group or the control group. The experimental group will accept group game-based activity twice a week lasting 12 weeks. There will be many motion-sensing games in the group game-based activities. The games designed for activities can provide somatosensory control including tactual, visual and auditory feedback. On the contrary, Participants in the control group will accept the activities the psychiatric day wards and halfway house offer as usual.

After 12 weeks, subjects in two groups will be asked to complete the first post-test questionnaire and physical examination(T2) which physiological values, physical ability, depression rating scale quality of life and motivation of group game-based activities will be included. Then, they will be asked to do the second post-test after 4 weeks without any intervention to investigate the long-term effect of the group game-based activities. The content of the questionnaire and physical examination will be the same as T2.

ELIGIBILITY:
Inclusion Criteria:

* Adults whose age is above 18
* Patients who diagnosed with schizophrenia spectrum disorders or bipolar disorders
* At present, you can go out, make friends, take care of your daily life, fully exercise your rights, and have full capacity as an adult, and have not been restricted by any legal declaration, so you do not need to obtain the consent of your legal representative to sign to participate in this study.

Exclusion Criteria:

* Those who have obvious limb movement disorders, such as congenital disability or hemiplegia after stroke, etc., which make them unable to participate in the group's game activities
* Those who are unwilling or unable to complete the signing of the written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Height | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Height in meters.
Ｗeight | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Weight in kilograms. Weighing machine will be used.
BMI | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Body Mass Index(BMI), Weight and height will be combined to report BMI in kg/m^2.
Ｗaist circumference | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  The measuring tape will pass through the middle point between the upper edge of the left and right intestinal bones and the lower edge of the ribs. The Length of the measuring tape will be the results of Ｗaist circumference.
Buttocks circumference | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  The measuring tape will pass through the high point of buttocks. The Length of the measuring tape will be the results of Ｗaist circumference.
10-meter walking time at comfortable | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Time in second. To measuring time of walking at comfortable for 10 meters.
10-meter walking time at maximum | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Time in second. Investigators will measure the time of walking at maximum for 10 meters.
Get up and Go test | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Time in second. First, The patient will sit on a chair. Second, he/she will stand up and go for 3 meters. At last, he/she will turn around and go back to have a sit. Investigators will measure time of the process.
5 times sit-to-stand-test | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Time in second. First, The patient will sit on a chair. Second, he/she will stand up and sit down immediately. The patients will be asked to do this process for 5 times.
Body fat percentage | T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16)
  Investigators will measure patients' body fat percentage by the body fat machine produced by Inbody company.

SECONDARY OUTCOMES:
Patient health questionnaire-9 | Depression rating scale will be done at T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16). motivation of group game-based activities will be at T2=first post-test(Week 12) and T3=second post-test(Week 16).
  The abbreviation of patient health questionnaire-9 is PHQ-9. The total number of questions is 9. The minimum and maximum values are 0 and 27 respectively. Then, the higher scores mean a worse outcome.
World Health Organization Quality-of-Life Scale | The questionnaire of quality of life will be done at T1=pre test, T2=first post-test(Week 12) and T3=second post-test(Week 16). motivation of group game-based activities will be at T2=first post-test(Week 12) and T3=second post-test(Week 16).
  The abbreviation of World Health Organization Quality-of-Life Scale is WHOQOL-BREF. The total number of questions is 28. The minimum and maximum values are 28 and 140 respectively. Then, the higher scores mean a better outcome.
Chinese version of interactive video games questionnaire on satisfaction and feasibility | Motivation of group game-based activities will be done at T2=first post-test(Week 12) and T3=second post-test(Week 16).
  The total number of questions is 13. The content of the questionnaire includes whether the games is easy, the games can bring happiness and deserve to play, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No